CLINICAL TRIAL: NCT04904276
Title: Observational Study of Fostamatinib as Second Line Therapy in Adult Patients With Immune Thrombocytopenia (ITP) and Insufficient Response to a Prior Therapy (FORTE)
Brief Title: Observational Study of Fostamatinib as Second Line Therapy in Adult Patients With Immune Thrombocytopenia (ITP) and Insufficient Response to a Prior Therapy
Status: Terminated | Type: Observational
Why Stopped: met minimum enrollment goal, however, enrollment was slow due to the pandemic, therefore, the study was terminated
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: O-FOSTA-901
Record Dates: First submitted 2021-04-13; First posted 2021-05-27 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: ITP; Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — fostamatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiating treatment with fostamatinib as second-line therapy
  Interventions: Drug: Fostamatinib
- Treated with fostamatinib for at least 12 weeks as second-line therapy
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib disodium

SUMMARY:
Evaluate patient characteristics, treatment patterns, clinical outcomes and safety of fostamatinib as second-line therapy in real-world clinical practice, for the treatment of ITP in adult patients who have an insufficient response to prior therapy (steroids ± immunoglobulins).

DETAILED DESCRIPTION:
Evaluate patient characteristics, treatment patterns, clinical outcomes and safety of fostamatinib as second-line therapy in real-world clinical practice, for the treatment of ITP in adult patients who have an insufficient response to prior therapy (steroids ± immunoglobulins).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Diagnosis of ITP in adult patients (≥ 18 years of age) with an insufficient response to steroids ± immunoglobulins and requiring a change in therapy
3. For Cohort 1, intent to initiate fostamatinib at enrollment as change in therapy
4. For Cohort 2, currently undergoing treatment with fostamatinib as second line therapy for at least 12 weeks, with the intent to continue, at the time of enrollment

Exclusion Criteria:

1. Any prior ITP therapy/treatment other than steroids ± immunoglobulins (e.g. rituximab, thrombopoietin receptor agonists (TPO), splenectomy)
2. Participation in any interventional study during the course of this study
3. Lack of historical platelet counts, at time of fostamatinib initiation for those entering Cohort 2
4. Pregnant and/or nursing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This two-cohort study will enroll approximately 45 patients diagnosed with ITP. Cohort 1 will enroll approximately 30 ITP patients who will begin treatment with fostamatinib as second-line therapy. Cohort 2 will enroll approximately 15 patients who have a record of at least 12 weeks of fostamatinib treatment as second-line therapy, with the intent to continue, at time of enrollment.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Fostamatinib dosing | 12-month observation period
  Changes in fostamatinib dosing
Platelet counts over time during the course of fostamatinib therapy | 12-month observation period
  Platelet count and change from baseline in platelet count over time.
Use of concomitant medications related to ITP | 12-month observation period
  Use of concomitant medications related to ITP during the study.
Use of ITP Rescue Medication | 12-month observation period
  The number of patients with ITP rescue medication use at any time during the study.
Safety of fostamatinib | 12-month observation period
  Evaluate continued safety of fostamatinib in ITP patients through adverse events
ITP-PAQ Quality of life measure | 12-month observation period
  Use of the score from questionnaire to assess disease-specific quality of life in adults with ITP.
Treatment satisfaction measure (MSQ) | 12-month observation period
SF-36 Quality of life measure | 12-month observation period
  Scale of functional health and well-being from the patient's point of view.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Advanced Research, Tamarac, Florida
  - Simmons Cancer Institute at Southern Illinois University, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Saint Agnes Hospital, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A, Clinton, Maryland
  - Maryland Oncology Hematology, P.A, Columbia, Maryland
  - Maryland Oncology Hematology, P.A, Rockville, Maryland
  - Maryland Oncology Hematology, P.A, Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Regional Cancer Care Associates, LLC, Little Silver, New Jersey
  - New York Medical College Westchester Medical Center, Valhalla, New York
  - New York Medical College, Valhalla, New York